CLINICAL TRIAL: NCT00561015
Title: A Phase IIa Randomized, Partially Blinded Trial of Telaprevir (VX-950) in Treatment-Naive Subjects With Chronic Genotype 2 or 3 Hepatitis C Infection
Brief Title: A Phase 2a Study to Evaluate Viral Kinetics and Safety of Telaprevir in Participants With Genotype 2 or 3 Hepatitis C Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec BVBA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR013513; VX-950-TiDP24-C209; NCT00613704 (obsolete NCT alias)
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Results first posted 2013-06-04 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C, Chronic; Genotype 2; Genotype 3; Telaprevir
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — telaprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- TVR then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 2 (Experimental): Participants who are never treated for chronic hepatitis C (inflammation of the liver) genotype 2 will receive telaprevir (TVR) 750 milligram (mg) tablet orally 3 times a day during investigational treatment phase from Day 1 to Day 15. Participants will then be treated with standard treatment regimen of pegylated interferon (Peg-IFN)-alfa-2a and ribavirin (RBV) from Day 15 to Week 26 (standard treatment phase). Each dose of pegylated interferon 180 microgram (mcg) will be administered as a subcutaneous injection once a week. RBV will be taken orally as 400 mg tablets 2 times a day. Total duration of treatment will be 26 weeks.
  Interventions: Drug: Telaprevir; Drug: Peg-IFN-alfa-2a + Ribavirin (Standard Treatment)
- TVR with Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 2 (Experimental): Participants who are never treated for CHC genotype 2 will receive TVR 750 mg tablet orally 3 times a day during investigational treatment phase from Day 1 to Day 15 along with standard treatment regimen of Peg-IFN-alfa-2a and RBV which will be continued in the standard treatment phase from Day 15 to Week 24. Each dose of Peg-IFN-alfa-2a 180 mcg will be administered as a subcutaneous injection once a week. RBV will be taken orally as 400 mg tablets 2 times a day. Total duration of treatment will be 24 weeks.
  Interventions: Drug: Telaprevir; Drug: Peg-IFN-alfa-2a + Ribavirin (Standard Treatment)
- Pbo with Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 2 (Active Comparator): Participants who are never treated for CHC genotype 2 will receive TVR matching placebo (Pbo) tablet orally 3 times a day during investigational treatment phase from Day 1 to Day 15 along with standard treatment regimen of Peg-IFN-alfa-2a and RBV which will be continued in the standard treatment phase from Day 15 to Week 24. Each dose of Peg-IFN-alfa-2a 180 mcg will be administered as a subcutaneous injection once a week. RBV will be taken orally as 400 mg tablets 2 times a day. Total duration of treatment will be 24 weeks.
  Interventions: Drug: Peg-IFN-alfa-2a + Ribavirin (Standard Treatment); Drug: Placebo
- TVR then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 3 (Experimental): Participants who are never treated for CHC genotype 3 will receive TVR 750 mg tablet orally 3 times a day during investigational treatment phase from Day 1 to Day 15. Participants will then be treated with standard treatment regimen of Peg-IFN-alfa-2a and RBV from Day 15 to Week 26 (standard treatment phase). Each dose of Peg-IFN-alfa-2a 180 mcg will be administered as a subcutaneous injection once a week. RBV will be taken orally as 400 mg tablets 2 times a day. Total duration of treatment will be 26 weeks.
  Interventions: Drug: Telaprevir; Drug: Peg-IFN-alfa-2a + Ribavirin (Standard Treatment)
- TVR with Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 3 (Experimental): Participants who are never treated for CHC genotype 3 received TVR 750 mg tablet orally 3 times a day during investigational treatment phase from Day 1 to Day 15 along with standard treatment regimen of Peg-IFN-alfa-2a and RBV which will be continued in the standard treatment phase from Day 15 to Week 24. Each dose of Peg-IFN-alfa-2a 180 mcg will be administered as a subcutaneous injection once a week. RBV will be taken orally as 400 mg tablets 2 times a day. Total duration of treatment will be 24 weeks.
  Interventions: Drug: Telaprevir; Drug: Peg-IFN-alfa-2a + Ribavirin (Standard Treatment)
- Pbo with Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 3 (Active Comparator): Participants who are never treated for CHC genotype 3 will receive TVR matching Pbo tablet orally 3 times a day during investigational treatment phase from Day 1 to Day 15 along with standard treatment regimen of Peg-IFN-alfa-2a and RBV which will be continued in the standard treatment phase from Day 15 to Week 24. Each dose of Peg-IFN-alfa-2a 180 mcg will be administered as a subcutaneous injection once a week. RBV will be taken orally as 400 mg tablets 2 times a day. Total duration of treatment will be 24 weeks.
  Interventions: Drug: Peg-IFN-alfa-2a + Ribavirin (Standard Treatment); Drug: Placebo

INTERVENTIONS:
Drug: Telaprevir — Telaprevir 750 mg tablet will be administered three times a day orally for 2 weeks.
  Other Names: VX-950
  Arms: TVR then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 2; TVR then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 3; TVR with Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 2; TVR with Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 3
Drug: Peg-IFN-alfa-2a + Ribavirin (Standard Treatment) — Standard treatment of Peg-IFN-alfa-2a (180 mcg subcutaneous injection, once weekly) and ribavirin (400 mg as oral tablet twice daily) will be administered from Day 15 to Week 24 or 26 in the T2 & PR24 - genotype 2 and 3 group and from Day 1 to Week 24 or 26 in the T2/PR24 - genotype 2 and 3 group.
Drug: Placebo — Matching placebo tablet to telaprevir will be administered three times a day orally for 2 weeks.
  Arms: Pbo with Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 2; Pbo with Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 3

SUMMARY:
The purpose of this study is to assess the effect of telaprevir on early hepatitis (inflammation of the liver) C virus (HCV) viral kinetics in treatment-naive participants who are chronically (lasting a long time) infected with genotype 2 or 3 HCV.

DETAILED DESCRIPTION:
This is a Phase 2a multicenter (when more than one hospital or medical school team work on a medical research study), partially blinded, randomized (study drug assigned by chance) stratified (arrange in groups for analysis of results e.g., stratify by age, sex, etc.) for genotype, multiple dose study. The trial will consist of Screening period (6 weeks), Treatment period (24 or 26 weeks) and Follow-up period (24 weeks). The Treatment period will include 2 weeks investigational treatment phase and a 24 week standard treatment phase. All the eligible participants who were never treated for HCV will be enrolled for the trial and will receive the investigational treatment regimen to which they have been randomly assigned for 2 weeks. After this in the standard treatment phase participants will receive the standard treatment of care consisting of pegylated interferon (Peg-IFN)-alfa-2a 180 microgram once weekly and ribavirin (RBV) 400 milligram twice per day. Efficacy will primarily be evaluated by HCV viral load quantification. Participant's safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants chronically infected with genotype 2 or 3 hepatitis C virus (HCV) with amount of virus in the blood greater than 10,000 international units per milliliter (IU/ml)
* Participants who were never treated for hepatitis C virus infection
* Participants without any significant lab abnormalities
* Participants who agree to the use of two effective methods of contraception
* Participant who were judged to be in good health

Exclusion Criteria:

* Participants who had contraindications for starting anti-HCV therapy
* Participants who had history or evidence of liver cirrhosis (serious liver disorder in which connective tissue replaces normal liver tissue, and liver failure often occurs) or decompensated liver disease or hepatocellular carcinoma (type of cancer)
* Participant infected with human immunodeficiency virus (a life-threatening infection that you can get from an infected person's blood or from having sex with an infected person) or hepatitis B virus
* Females who are pregnant (carrying an unborn baby), planning to be pregnant or breastfeeding
* Participants who have hypersensitivity to tartrazine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec-Virco Virology BVBA Clinical Trial, Study Director — Tibotec BVBA
Locations (7):
- France (5):
  - Clichy
  - Créteil
  - Lyon
  - Paris
  - Vandœuvre-lès-Nancy
- Stockholm, Sweden
- London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 26 participants infected with genotype 2 hepatitis C virus (HCV) who were randomly assigned to treatment, only 23 participants received treatment. 2 participants withdrew and 1 participant was infected with HCV genotype 4. All the 26 participants infected with genotype 3 HCV received treatment.
Groups:
- TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 2: Participants who were never treated for chronic hepatitis (inflammation of liver) C genotype 2 received telaprevir (TVR) 750 milligram (mg) tablet orally 3 times a day during investigational treatment phase from Day 1 to Day 15. Participants were then treated with standard treatment regimen of pegylated interferon (Peg-IFN)-alfa-2a and ribavirin (RBV) from Day 15 to Week 26 (standard treatment phase). Each dose of Peg-IFN-alfa-2a 180 microgram (mcg) was administered as a subcutaneous injection once a week. RBV was taken orally as 400 mg tablets 2 times a day. Total duration of treatment was 26 weeks.
- TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 2: Participants who were never treated for chronic hepatitis C genotype 2 received TVR 750 mg tablet orally 3 times a day during investigational treatment phase from Day 1 to Day 15 along with standard treatment regimen of Peg-IFN-alfa-2a and RBV which was continued in the standard treatment phase from Day 15 to Week 24. Each dose of Peg-IFN-alfa-2a 180 mcg was administered as a subcutaneous injection once a week. RBV was taken orally as 400 mg tablets 2 times a day. Total duration of treatment was 24 weeks.
- Pbo With Peg-IFN-alfa-2a+ RBV (Pbo/PR24) - Genotype 2: Participants who were never treated for chronic hepatitis C genotype 2 received TVR matching placebo (Pbo) tablet orally 3 times a day during investigational treatment phase from Day 1 to Day 15 along with standard treatment regimen of Peg-IFN-alfa-2a and RBV which was continued in the standard treatment phase from Day 15 to Week 24. Each dose of Peg-IFN-alfa-2a 180 mcg was administered as a subcutaneous injection once a week. RBV was taken orally as 400 mg tablets 2 times a day. Total duration of treatment was 24 weeks.
- TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 3: Participants who were never treated for chronic hepatitis C genotype 3 received TVR 750 mg tablet orally 3 times a day during investigational treatment phase from Day 1 to Day 15. Participants were then treated with standard treatment regimen of Peg-IFN-alfa-2a and RBV from Day 15 to Week 26 (standard treatment phase). Each dose of Peg-IFN-alfa-2a 180 mcg was administered as a subcutaneous injection once a week. RBV was taken orally as 400 mg tablets 2 times a day. Total duration of treatment was 26 weeks.
- TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 3: Participants who were never treated for chronic hepatitis C genotype 3 received TVR 750 mg tablet orally 3 times a day during investigational treatment phase from Day 1 to Day 15 along with standard treatment regimen of Peg-IFN-alfa-2a and RBV which was continued in the standard treatment phase from Day 15 to Week 24. Each dose of Peg-IFN-alfa-2a 180 mcg was administered as a subcutaneous injection once a week. RBV was taken orally as 400 mg tablets 2 times a day. Total duration of treatment was 24 weeks.
- Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 3: Participants who were never treated for chronic hepatitis C genotype 3 received TVR matching Pbo tablet orally 3 times a day during investigational treatment phase from Day 1 to Day 15 along with standard treatment regimen of Peg-IFN-alfa-2a and RBV which was continued in the standard treatment phase from Day 15 to Week 24. Each dose of Peg-IFN-alfa-2a 180 mcg was administered as a subcutaneous injection once a week. RBV was taken orally as 400 mg tablets 2 times a day. Total duration of treatment was 24 weeks.
Period: Overall Study
Arm/Group | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 2 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 2 | Pbo With Peg-IFN-alfa-2a+ RBV (Pbo/PR24) - Genotype 2 | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 3 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 3 | Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 3
Started | 9 | 5 | 9 | 8 | 9 | 9
Completed | 5 | 5 | 9 | 7 | 8 | 6
Not Completed | 4 | 0 | 0 | 1 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 1 | 0 | 3
Not completed — Participant non-compliance | 2 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 2: Participants who were never treated for chronic hepatitis C genotype 2 received telaprevir (TVR) 750 milligram (mg) tablet orally 3 times a day during investigational treatment phase from Day 1 to Day 15. Participants were then treated with standard treatment regimen of pegylated interferon (Peg-IFN)-alfa-2a and ribavirin (RBV) from Day 15 to Week 26 (standard treatment phase). Each dose of Peg-IFN-alfa-2a 180 microgram (mcg) was administered as a subcutaneous injection once a week. RBV was taken orally as 400 mg tablets 2 times a day. Total duration of treatment was 26 weeks.
- Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 2: Participants who were never treated for CHC genotype 2 received TVR matching placebo (Pbo) tablet orally 3 times a day during investigational treatment phase from Day 1 to Day 15 along with standard treatment regimen of Peg-IFN-alfa-2a and RBV which was continued in the standard treatment phase from Day 15 to Week 24. Each dose of Peg-IFN-alfa-2a 180 mcg was administered as a subcutaneous injection once a week. RBV was taken orally as 400 mg tablets 2 times a day. Total duration of treatment was 24 weeks.
- Total: Total of all reporting groups
Arm/Group | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 2 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 2 | Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 2 | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 3 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 3 | Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 3 | Total
Number analyzed (Participants) | 9 | 5 | 9 | 8 | 9 | 9 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 5 | 9 | 8 | 9 | 9 | 49
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 42.3 (10.63) | 56.6 (5.13) | 49.8 (10.33) | 43.4 (9.62) | 42.4 (7.75) | 39.8 (13.76) | 44.9 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 4 | 3 | 1 | 0 | 14
  Male | 7 | 1 | 5 | 5 | 8 | 9 | 35
Region of Enrollment [Number; unit: participants]
  France | 7 | 5 | 6 | 3 | 4 | 3 | 28
  Italy | 1 | 0 | 2 | 0 | 0 | 1 | 4
  Sweden | 0 | 0 | 1 | 0 | 0 | 0 | 1
  United Kingdom | 1 | 0 | 0 | 5 | 5 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Log 10 Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Level at Day 15
Description: Level of HCV RNA in plasma was measured using COBAS TaqMan HCV test v2.0 (an in vitro nucleic acid amplification test for quantitation of HCV RNA genotypes 1 through 6 in human serum or plasma, using the COBAS AmpliPrep Total Nucleic Acid Isolation Kit (TNAI) for preparation of highly purified total nucleic acid from serum or plasma and automated amplification and detection on TaqMan 48 Analyzer). Lower limit of quantification was 25 international units/milliliter (IU/ml) and limit of detection was 10 IU/ml. Assay used was reverse transcription-polymerase chain reaction (RT-PCR) methodology.
Time Frame: Baseline, Pre-dose (Day 15)
Population: Full analysis set (FAS) population included all randomly assigned participants who received at least 1 dose of TVR or placebo.
Measure: Median (Full Range); unit: log10 IU/ml
Arm/Group | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 2 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 2 | Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 2 | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 3 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 3 | Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 3
Number analyzed (Participants) | 9 | 5 | 9 | 8 | 9 | 9
log10 IU/ml
  Baseline | 6.61 [4.4 to 7.3] | 6.21 [5.3 to 7.3] | 6.15 [5.5 to 7.4] | 6.65 [5.8 to 7.1] | 6.79 [5.4 to 7.4] | 6.92 [3.9 to 7.3]
  Change at Day 15 | -3.66 [-5.4 to -0.9] | -5.51 [-6.0 to -4.6] | -4.83 [-6.0 to -0.2] | -0.54 [-1.0 to -0.1] | -4.85 [-6.1 to -2.3] | -4.72 [-6.1 to -3.2]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) for Telaprevir on Day 1
Description: The Cmax is defined as the maximum observed analyte concentration. The Cmax was measured in nanogram/milliliter (ng/ml).
Time Frame: Pre-dose Day 1 (0.5, 1, 2, 3, 4, 6, 8 hour [hr])
Population: The FAS population included all randomly assigned participants who received at least 1 dose of TVR or placebo. Here 'N' (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- TVR With Peg-IFN-alfa-2a on + RBV (T2/PR24) - Genotype 3: Participants who were never treated for CHC genotype 3 received TVR 750 mg tablet orally 3 times a day during investigational treatment phase from Day 1 to Day 15 along with standard treatment regimen of Peg-IFN-alfa-2a and RBV which was continued in the standard treatment phase from Day 15 to Week 24. Each dose of Peg-IFN-alfa-2a 180 mcg was administered as a subcutaneous injection once a week. RBV was taken orally as 400 mg tablets 2 times a day. Total duration of treatment was 24 weeks.
Arm/Group | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 2 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 2 | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 3 | TVR With Peg-IFN-alfa-2a on + RBV (T2/PR24) - Genotype 3
Number analyzed (Participants) | 9 | 5 | 7 | 8
ng/ml | 1886 (1043) | 2462 (761) | 1497 (435) | 1588 (1090)

3. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) for Telaprevir on Day 1
Description: The Tmax is defined as the actual sampling time to reach maximum observed analyte concentration. The analyte concentration associated with Tmax is referred to as Cmax.
Time Frame: Pre-dose Day 1 (0.5, 1, 2, 3, 4, 6, 8 hr)
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 2 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 2 | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 3 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 3
Number analyzed (Participants) | 9 | 5 | 7 | 8
hr | 3.0 [0.5 to 6.0] | 4.0 [2.1 to 4.2] | 4.0 [3.0 to 6.0] | 4.0 [3.0 to 8.0]

4. Secondary Outcome: Area Under Plasma Concentration-Time Curve Over Dosing Interval (AUCtau) for Telaprevir on Day 15
Description: The AUC is defined as area under the plasma concentration-time curve over the dosing interval (8 hr), calculated by the lin-up/ log-down method.
Time Frame: Pre-dose Day 15 (0.5, 1, 2, 3, 4, 6, 8 hr)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 2 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 2 | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 3 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 3
Number analyzed (Participants) | 8 | 4 | 6 | 6
ng*hr/ml | 20144 (11129) | 26588 (10908) | 18480 (3011) | 20895 (6242)

5. Secondary Outcome: Change From Baseline in Log 10 Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Level at Week 24 and Week 26
Description: Levels of HCV RNA in plasma were measured using COBAS TaqMan HCV test v2.0. Lower limit of quantification was 25 IU/ml and limit of detection was 10 IU/ml. The assay used real time RT-PCR methodology. End of treatment (EOT) for group T2 & PR24 was 26 weeks and for groups T2/PR24 and Pbo/PR24 was 24 weeks.
Time Frame: Baseline and Week 24/26
Population: as for outcome 2
Measure: Median (Full Range); unit: log10 IU/ml
Groups:
- Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 2: Participants who were never treated for CHC genotype 2 received TVR matching Pbo tablet orally 3 times a day during investigational treatment phase from Day 1 to Day 15 along with standard treatment regimen of Peg-IFN-alfa-2a and RBV which was continued in the standard treatment phase from Day 15 to Week 24. Each dose of Peg-IFN-alfa-2a 180 mcg was administered as a subcutaneous injection once a week. RBV was taken orally as 400 mg tablets 2 times a day. Total duration of treatment was 24 weeks.
Arm/Group | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 2 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 2 | Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 2 | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 3 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 3 | Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 3
Number analyzed (Participants) | 7 | 5 | 9 | 8 | 7 | 9
log10 IU/ml | -5.91 [-6.6 to -3.7] | -5.51 [-6.6 to -4.6] | -5.45 [-6.7 to 0.7] | -5.71 [-6.4 to -0.9] | -5.50 [-6.7 to -4.7] | -6.22 [-6.6 to -3.2]

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) for Telaprevir on Day 15
Description: The Cmax is defined as the maximum observed analyte concentration. The Cmax is measured in ng/ml.
Time Frame: Pre-dose Day 15 (0.5, 1, 2, 3, 4, 6, 8 hr)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 2 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 2 | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 3 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 3
Number analyzed (Participants) | 8 | 4 | 6 | 6
ng/ml | 3261 (1818) | 4318 (1518) | 2898 (423) | 3358 (377)

7. Secondary Outcome: Minimum Plasma Concentration (Cmin) for Telaprevir on Day 15
Description: The Cmin is defined as minimum plasma concentration between 0 hr and dosing interval. The Cmin is measured in ng/ml.
Time Frame: Pre-dose Day 15 (0.5, 1, 2, 3, 4, 6, 8 hr)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 2 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 2 | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 3 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 3
Number analyzed (Participants) | 8 | 4 | 6 | 6
ng/ml | 1605 (1106) | 2164 (1398) | 1800 (375) | 2002 (659)

8. Primary Outcome: Area Under Plasma Concentration-Time Curve Over Dosing Interval (AUCtau) for Telaprevir on Day 1
Description: as for outcome 4
Time Frame: Pre-dose Day 1 (0.5, 1, 2, 3, 4, 6, 8 hr)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 2 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 2 | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 3 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 3
Number analyzed (Participants) | 9 | 5 | 7 | 8
ng*hr/ml | 7980 (4658) | 11248 (3810) | 6938 (1828) | 6979 (5011)

9. Secondary Outcome: Percentage of Participants Achieving Virological Response (HCV RNA Level < 10 IU/ml)
Description: Virological response was defined as having HCV RNA level less than a particular threshold that is less than 10 IU/ml (undetectable).
Time Frame: Baseline, Day 12, 15, Week 4, 6, 14 and EOT (Week 24/26 or early discontinuation)
Population: The FAS population included all randomly assigned participants who received at least 1 dose of TVR or placebo. Here 'n' included those participants who were evaluable for this measure at specific time points.
Measure: Number; unit: percentage of participants
Arm/Group | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 2 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 2 | Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 2 | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 3 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 3 | Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 3
Number analyzed (Participants) | 9 | 5 | 9 | 8 | 9 | 9
percentage of participants
  Day 12 (n=8,5,9,8,9,9) | 0.00 | 60.0 | 0.00 | 0.00 | 11.1 | 22.2
  Day 15 (n=9,5,9,8,9,9) | 0.00 | 40.0 | 22.2 | 0.00 | 22.2 | 11.1
  Week 4 (n=7,5,9,8,9,9) | 71.4 | 80.0 | 44.4 | 0.00 | 33.3 | 66.7
  Week 6 (n=7,5,9,8,9,9) | 71.4 | 100.0 | 77.8 | 37.5 | 66.7 | 100
  Week 14 (n=7,5,9,8,9,9) | 100 | 100.0 | 88.9 | 75.0 | 100 | 100
  Week 24/ Week 26 (n=7,5,9,8,7,9) | 100 | 100.0 | 88.9 | 75.0 | 100 | 100
  EOT (n=9,5,9,8,9,9) | 88.9 | 100.0 | 88.9 | 75.0 | 100 | 100

10. Secondary Outcome: Median Time to Virological Response (HCV RNA Level < 10 IU/ml)
Description: Virological response was defined as having HCV RNA level less than a particular threshold which is either less than 10 IU/ml (undetectable) or less than 25 IU/ml (unquantifiable).Time to virological response was defined as the number of days from the start of medication intake necessary to go for the first time below the threshold value. The EOT for group T2 & PR24 was 26 weeks and for groups T2/PR24 and Pbo/PR24 was 24 weeks.
Time Frame: Baseline up to EOT
Population: The FAS population included all randomly assigned participants who received at least 1 dose of TVR or placebo.
Measure: Median (Full Range); unit: days
Arm/Group | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 2 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 2 | Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 2 | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 3 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 3 | Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 3
Number analyzed (Participants) | 9 | 5 | 9 | 8 | 9 | 9
days | 31.0 [29.0 to 45.0] | 12.0 [8.0 to 29.0] | 43.0 [29.0 to 45.0] | 99.0 [46.0 to 185.0] | 43.0 [15.0 to 99.0] | 29.0 [29.0 to 39.0]

11. Secondary Outcome: Percentage of Participants With Viral Breakthrough
Description: Viral breakthrough was defined as an increase in HCV RNA levels by more than 1 log10 in HCV RNA level from the lowest level reached, or a value of HCV RNA > 100 IU/ml in participants whose HCV RNA had previously become undetectable (< 10 IU/ml) or unquantifiable (< 25 IU/ml) during the considered treatment phase. It was considered as confirmed when the criterion for viral breakthrough is fulfilled at two or more consecutive time points or at the last observed time point in case of trial termination. The EOT for group T2 & PR24 was 26 weeks and for groups T2/PR24 and Pbo/PR24 was 24 weeks.
Time Frame: Baseline, Day 12, 15 and Week 24/26
Population: The FAS population included all randomly assigned participants who received at least 1 dose of TVR or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 2 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 2 | Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 2 | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 3 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 3 | Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 3
Number analyzed (Participants) | 9 | 5 | 9 | 8 | 9 | 9
percentage of participants
  Day 12 | 11.1 | 0.0 | 0.0 | 37.5 | 0.0 | 0.0
  Day 15 | 66.7 | 0.0 | 0.0 | 37.5 | 0.0 | 0.0
  Week 24/ Week 26 | 66.7 | 0.0 | 11.1 | 37.5 | 0.0 | 0.0

12. Secondary Outcome: Percentage of Participants Who Demonstrated Virological Relapse
Description: Relapse was defined as confirmed detectable HCV RNA (>=10 IU/ml) during the follow-up period up to 24 weeks after last medication intake and after previous undetectable HCV RNA (< 10 IU/ml) at EOT. No relapse was defined as having no confirmed detectable HCV RNA (>=10 IU/ml) during the follow-up period and after previous undetectable HCV RNA (< 10 IU/ml) at EOT. Missing follow-up means no HCV RNA measurements during the follow-up period and after previous undetectable HCV RNA (< 10 IU/ml) at EOT. The EOT for group T2 & PR24 was 26 weeks and for groups T2/PR24 and Pbo/PR24 was 24 weeks.
Time Frame: 24 weeks after EOT
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 2 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 2 | Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 2 | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 3 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 3 | Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 3
Number analyzed (Participants) | 8 | 5 | 8 | 6 | 9 | 9
percentage of participants
  24 weeks after EOT | 12.5 | 0.0 | 0.0 | 33.3 | 33.3 | 22.2
  Missing follow-up | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 11.1

13. Secondary Outcome: Percentage of Participants Who Achieved Sustained Virological Response (SVR)
Description: The SVR was defined as having HCV RNA undetectable at EOT, not showing relapse up to follow-up Week 12 (SVR12) or follow-up Week 24 (SVR24), and HCV RNA undetectable at follow-up Week 12 (SVR12) or follow-up Week 24 (SVR24), respectively. The EOT for group T2 & PR24 was 26 weeks and for groups T2/PR24 and Pbo/PR24 was 24 weeks.
Time Frame: Week 12, 24 after EOT
Population: The FAS population included all randomly assigned participants who received at least 1 dose of TVR or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 2 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 2 | Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 2 | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 3 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 3 | Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 3
Number analyzed (Participants) | 9 | 5 | 9 | 8 | 9 | 9
percentage of participants
  SVR 12 | 66.7 | 100 | 88.9 | 50.0 | 66.7 | 44.4
  SVR 24 | 55.6 | 100 | 88.9 | 50.0 | 66.7 | 44.4

ADVERSE EVENTS:
Time Frame: Screening period (Week minus 6) up to 2 weeks of telaprevir treatment phase.
Groups:
- Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 2: Participants who were never treated for CHC genotype 2 received TVR matching placebo (Pbo) tablet orally 3 times a day during investigational treatment phase from Day 1 to Day 15 along with standard treatment regimen of Peg-IFN-alfa-2a and RBV which was continued in the standard treatment phase from Day 15 to Week 24. Each dose of Peg-IFN-alfa-2a180 mcg was administered as a subcutaneous injection once a week. RBV was taken orally as 400 mg tablets 2 times a day. Total duration of treatment was 24 weeks.
Arm/Group | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 2 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 2 | Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 2 | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 3 | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 3 | Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 3
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/5 | 0/9 | 0/8 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 6/9 | 4/5 | 8/9 | 7/8 | 9/9 | 8/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 2 (N=9) | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 2 (N=5) | Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 2 (N=9) | TVR Then Peg-IFN-alfa-2a + RBV (T2 & PR24) - Genotype 3 (N=8) | TVR With Peg-IFN-alfa-2a + RBV (T2/PR24) - Genotype 3 (N=9) | Pbo With Peg-IFN-alfa-2a + RBV (Pbo/PR24) - Genotype 3 (N=9)
Asthenia (General disorders) | 4 | 2 | 3 | 1 | 2 | 2
Influenza like illness (General disorders) | 1 | 2 | 3 | 3 | 5 | 4
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 1 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 4 | 1
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Irritability (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 2 | 0 | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 4 | 1 | 2 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 2 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 1 | 0 | 4 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 2 | 0
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 3 | 2 | 1 | 3
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Parosmia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
As per revised Protocol dated 14 Feb 2008, Investigator may not submit for publication or presentation, the results of trial without prior written consent of Sponsor. The Investigator agrees to allow at least 45 days for Sponsor to review pre-publication manuscript prior to submission to Publisher. In accordance with generally recognized principles of scientific collaboration, co-authorship with any company personnel will be discussed and mutually agreed upon before submission to Publisher.